CLINICAL TRIAL: NCT02196337
Title: Salt Iodization and the 1st 1000 Days: Does a USI Program Cover the Iodine Requirement of Pregnant and Lactating Women and Infants?
Brief Title: Salt Iodization: Meeting the Needs of Pregnancy, Lactation and Infancy
Acronym: SIMPLIFY
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zagreb (Other); St. Luke's Medical Center (Other); Global Alliance for Improved Nutrition (Other); UNICEF (Other); Shanxi Institute for Prevention and Treatment of Endemic Disease (Unknown)
Responsible Party: Principal Investigator, Maria Andersson, PhD, Swiss Federal Institute of Technology
Other Study IDs: EK 2013-N-82
Record Dates: First submitted 2014-06-02; First posted 2014-07-22 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Iodine Deficiency
Keywords: Iodine deficiency

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine, dried blood spots, breast milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Women of reproductive age: Age: 18-44 years
- Pregnant women: Age: 18-44 years
- Lactating women: Age: 18-44 years
- Young infants: Age: younger than 6 months
- Toddlers: Age: between 6 and 24 months
- School-aged children: Age: 6-12 years

SUMMARY:
The purpose of this study is to determine whether universal salt iodization (USI) meets the iodine requirements of pregnant women, lactating women and infants.

DETAILED DESCRIPTION:
Because pregnant women, lactating women and infants are the groups most vulnerable to iodine deficiency and its irreversible consequences, programs should focus on these groups. But like other mass fortification strategies, it is uncertain whether USI can meet the increased dietary requirements of pregnant women, lactating women and infants. Objective of this study to test whether USI can meet the dietary requirements of iodine in women of reproductive age, pregnant women, lactating women and infants up to 2 years of age without causing excess iodine intake in school children and non-pregnant non-lactating women. The study hypothesis is that USI, when fortified at adequate levels and applied to all salt consumed, including both household salt and salt used for processed foods, provides adequate dietary iodine for all population groups, except for weaning infants; while not posing any risk of excessive iodine intakes in other age groups.

ELIGIBILITY:
Inclusion Criteria:

* living at study area for at least 6 months
* generally healthy
* no chronic medication
* no history of thyroid disease in the family
* no use of iodine containing dietary supplements during the last 6 months
* no use of iodine containing disinfectants for the last 6 months
* no use of X-ray / CT contrast agent or iodine containing medication within the last year
* in addition for women of reproductive age, pregnant women and breastfeeding women: age between 18 and 44 years old
* in addition for pregnant women: healthy pregnancy, singleton pregnancy (no twins or multiple pregnancy)
* in addition for breastfeeding women and breastfed infants: healthy pregnancy, singleton pregnancy (no twins or multiple pregnancy), baby born at full-term (in pregnancy week 38 to 42), the baby had normal birth weight (≥ 2500 g), baby not older than 6 months, baby currently completely breastfed (except for water, tea and juices)
* in addition for toddlers: between 6 and 24 months old

Ages: 2 Weeks to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In each of the four study countries, six population groups will be studied:
  * women of reproductive age
  * pregnant women
  * lactating women
  * young infants
  * toddlers
  * school-aged children
Sampling Method: Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration (µg/L) | 1 day
  Participants will be assessed only once. However, for 30% of the study participants urinary iodine concentration will be assessed in spot samples collected on two different days, spread over an expected average of 5 days.

SECONDARY OUTCOMES:
Thyroglobulin (µg/L) | 1 day
  Thyroglobulin will be measured in all population groups
Breast milk iodine concentration (µg/L) | 1 day
  Breast milk iodine concentration will be measured in lactating women.

OTHER OUTCOMES:
Thyroid function (TSH, T4) | 1 day
  Thyroid function (TSH, T4) will be measured where relevant.
Urinary sodium excretion (mg/day) | 1 day
  Urinary sodium excretion will be assessed in school age children and women of reproductive age. Participants will be assessed only once. However, for urinary sodium excretion 30% of the study participants will be assessed in spot samples collected on two different days, spread over an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria Andersson, PhD, Principal Investigator — ETH Zurich
Locations (4):
- Shanxi Institute for Prevention and Treatment of Endemic Disease, Linfen, Shanxi, China
- University of Zagreb, Zagreb, Croatia
- University of Santo Tomas Hospital, Manila, Philippines
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dold S, Zimmermann MB, Jukic T, Kusic Z, Jia Q, Sang Z, Quirino A, San Luis TOL, Fingerhut R, Kupka R, Timmer A, Garrett GS, Andersson M. Universal Salt Iodization Provides Sufficient Dietary Iodine to Achieve Adequate Iodine Nutrition during the First 1000 Days: A Cross-Sectional Multicenter Study. J Nutr. 2018 Apr 1;148(4):587-598. doi: 10.1093/jn/nxy015. PMID 29659964
- [Derived] Dold S, Zimmermann MB, Aboussad A, Cherkaoui M, Jia Q, Jukic T, Kusic Z, Quirino A, Sang Z, San Luis TO, Vandea E, Andersson M. Breast Milk Iodine Concentration Is a More Accurate Biomarker of Iodine Status Than Urinary Iodine Concentration in Exclusively Breastfeeding Women. J Nutr. 2017 Apr;147(4):528-537. doi: 10.3945/jn.116.242560. Epub 2017 Feb 22. PMID 28228508